CLINICAL TRIAL: NCT00825825
Title: A Comparison of the CNS Effects of Equivalent Doses of Escitalopram and Racemic Citalopram Using BOLD fMRI
Brief Title: Brain Effects of Escitalopram and Citalopram Using fMRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Henry, MD (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Michael Henry, MD, Principal Investigator, Steward St. Elizabeth's Medical Center of Boston, Inc.
Organization: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 00397
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Antidepressant Activity in Healthy Volunteers
Keywords: Citalopram; Escitalopram; Celexa; Lexapro; fMRI; antidepressant; healthy volunteers
MeSH Terms: interventions — Escitalopram; Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Escitalopram (Active Comparator): One week of escitalopram at 10 mg followed by one week at 20 mg in healthy volunteers.
  Interventions: Drug: Escitalopram
- Citalopram (Active Comparator): One week of citalopram at 20 mg followed by one week at 40 mg in healthy volunteers.
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Two weeks of placebo in healthy volunteers.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — One week of escitalopram taken orally at 10 mg followed by one week at 20 mg daily.
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Citalopram — One week of citalopram taken orally at 20 mg followed by one week at 40 mg daily.
  Other Names: Celexa
  Arms: Citalopram
Drug: Placebo — Two weeks of placebo taken orally.
  Arms: Placebo

SUMMARY:
Escitalopram (Lexapro) and citalopram (Celexa) are similar selective serotonin reuptake inhibitors that alter blood flow to the amygdala and other brain structures involved in regulating mood. Escitalopram consists of S-citalopram while citalopram contains both S-citalopram and R-citalopram (racemic citalopram). There is evidence that R-citalopram may block the effects of S-citalopram. The hypothesis being tested is that because of the antagonist effect of R-citalopram, S-citalopram will have a greater effect on the mood circuit than racemic citalopram when equal doses of S-citalopram are administered. The study design consists of a two week medication period followed by blood oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) while viewing affective visual stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 21 to 50 years.
* Capable of providing informed consent.
* Has an established residence and phone.

Exclusion Criteria:

* Meets DSM-IV criteria for an Axis I or II disorder.
* History of substance dependence or abuse within the past month.
* Use of NSAID's, beta blockers, calcium channel blockers, antidepressants, antipsychotic medications, lithium or other medication which in the opinion of the investigator would alter vascular responsivity.
* Regular use of sedative hypnotic or narcotic medication, or other medication that might affect the individual's perception of visual stimuli.
* History of cataracts or significant visual impairment.
* A medical condition, which in the opinion of the investigator is likely to affect the individual's perception of the visual stimuli or vascular response.
* Participation in a research protocol that included administration of medication within the past 3 months.
* Cigarette smoking.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Henry, MD, Principal Investigator — Steward St. Elizabeth's Medical Center
Locations (1):
- Steward St. Elizabeth's Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Windischberger C, Lanzenberger R, Holik A, Spindelegger C, Stein P, Moser U, Gerstl F, Fink M, Moser E, Kasper S. Area-specific modulation of neural activation comparing escitalopram and citalopram revealed by pharmaco-fMRI: a randomized cross-over study. Neuroimage. 2010 Jan 15;49(2):1161-70. doi: 10.1016/j.neuroimage.2009.10.013. Epub 2009 Oct 13. PMID 19833214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by advertisement from April 2008 until January 2011.
Pre-assignment Details: Participants had their serotonin transporter genotyped. Individuals with a genotype of SS or SLg were not randomized. A total of 85 potential participants were screened. Of those, 21 were excluded on the basis of genotype. Another 28 were determined to be ineligible for other reasons and 6 withdrew prior to randomization.
Groups:
- Escitalopram First / Citalopram Second / Placebo Third: 2 weeks of escitalopram followed by 2 weeks of citalopram followed by 2 weeks of placebo
- Escitalopram First / Placebo Second / Citalopram Third: 2 weeks of escitalopram followed by 2 weeks of placebo followed by 2 weeks of citalopram
- Citalopram First / Escitalopram Second / Placebo Third: 2 weeks of citalopram followed by 2 weeks of escitalopram followed by 2 weeks of placebo
- Citalopram First / Placebo Second / Escitalopram Third: 2 weeks of citalopram followed by 2 weeks of placebo followed by 2 weeks of escitalopram
- Placebo First / Escitalopram Second / Citalopram Third: 2 weeks of placebo followed by 2 weeks of escitalopram followed by 2 weeks of citalopram
- Placebo First / Citalopram Second / Escitalopram Third: 2 weeks of placebo followed by 2 weeks of citalopram followed by 2 weeks escitalopram
Period: First Medication Period (14 Days)
Arm/Group | Escitalopram First / Citalopram Second / Placebo Third | Escitalopram First / Placebo Second / Citalopram Third | Citalopram First / Escitalopram Second / Placebo Third | Citalopram First / Placebo Second / Escitalopram Third | Placebo First / Escitalopram Second / Citalopram Third | Placebo First / Citalopram Second / Escitalopram Third
Started | 6 | 4 | 3 | 5 | 4 | 5
Completed | 3 | 4 | 2 | 5 | 4 | 3
Not Completed | 3 | 0 | 1 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 1 | 0 | 0 | 1
Period: First Washout Period (14 Days)
Arm/Group | Escitalopram First / Citalopram Second / Placebo Third | Escitalopram First / Placebo Second / Citalopram Third | Citalopram First / Escitalopram Second / Placebo Third | Citalopram First / Placebo Second / Escitalopram Third | Placebo First / Escitalopram Second / Citalopram Third | Placebo First / Citalopram Second / Escitalopram Third
Started | 3 | 4 | 2 | 5 | 4 | 3
Completed | 3 | 4 | 2 | 5 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Medication Period (14 Days)
Arm/Group | Escitalopram First / Citalopram Second / Placebo Third | Escitalopram First / Placebo Second / Citalopram Third | Citalopram First / Escitalopram Second / Placebo Third | Citalopram First / Placebo Second / Escitalopram Third | Placebo First / Escitalopram Second / Citalopram Third | Placebo First / Citalopram Second / Escitalopram Third
Started | 3 | 4 | 2 | 5 | 4 | 3
Completed | 1 | 4 | 2 | 3 | 3 | 3
Not Completed | 2 | 0 | 0 | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1 | 0
Period: Second Washout Period (14 Days)
Arm/Group | Escitalopram First / Citalopram Second / Placebo Third | Escitalopram First / Placebo Second / Citalopram Third | Citalopram First / Escitalopram Second / Placebo Third | Citalopram First / Placebo Second / Escitalopram Third | Placebo First / Escitalopram Second / Citalopram Third | Placebo First / Citalopram Second / Escitalopram Third
Started | 1 | 4 | 2 | 3 | 3 | 3
Completed | 1 | 4 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Medication Period (14 Days)
Arm/Group | Escitalopram First / Citalopram Second / Placebo Third | Escitalopram First / Placebo Second / Citalopram Third | Citalopram First / Escitalopram Second / Placebo Third | Citalopram First / Placebo Second / Escitalopram Third | Placebo First / Escitalopram Second / Citalopram Third | Placebo First / Citalopram Second / Escitalopram Third
Started | 1 | 4 | 2 | 3 | 3 | 3
Completed | 1 | 2 | 2 | 3 | 3 | 1
Not Completed | 0 | 2 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 2
Not completed — poor data quality | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all randomized subjects regardless of order in which they received medications
Arm/Group | Entire Study Population
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Voxels Showing Greater Activation Following Escitalopram Compared With Citalopram When Happy and Fearful Faces Are Presented in a Rapid Covert Stimulus Presentation.
Description: Activation was measured using BOLD fMRI in response to happy and fearful faces presented in a rapid covert or masked presentation. The response following two weeks of escitalopram was compared to the response following two weeks of citalopram. The cluster of differential activation was located in the left middle temporal gyrus.
Time Frame: two weeks
Population: Participants were only included in the analysis if they had complete data for all 3 fMRI scans and motion was within acceptable limits. Participants also had to have detectable plasma levels of R-citalopram and S-citalopram in order to be included in the final analysis.
Measure: Number; unit: voxels
Groups:
- All Participants With Complete Usable Data: Participants were healthy volunteers who completed three medication periods of two weeks each (escitalopram, citalopram, and placebo) and had a successful magnetic resonance scan at the end of each medication period. The study design was a randomized crossover trial so all individuals received all interventions.
Arm/Group | All Participants With Complete Usable Data
Number analyzed (Participants) | 11
voxels | 478
Statistical Analysis 1: Comparison: All Participants With Complete Usable Data; This analysis is a comparison between the escitalopram and citalopram medication periods; Test type: Superiority or Other; p = 0.000704, Mixed Models Analysis

2. Secondary Outcome: Number of Voxels Showing Greater Activation Following Escitalopram Compared With Citalopram When Faces and a Fixation Stimulus Are Presented in an Overt Presentation.
Description: Activation was measured using BOLD fMRI in response to affective faces and a fixation stimulus presented in an overt or unmasked presentation. The response following two weeks of escitalopram was compared to the response following two weeks of citalopram. The cluster of differential activation was located in the right insular cortex.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Number; unit: voxels
Groups:
- All Participants With Complete Usuable Data: Participants were healthy volunteers who completed three medication periods of two weeks each (escitalopram, citalopram, and placebo) and had a successful magnetic resonance scan at the end of each medication period. The study design was a randomized crossover trial so all individuals received all interventions.
Arm/Group | All Participants With Complete Usuable Data
Number analyzed (Participants) | 11
voxels | 735
Statistical Analysis 1: Comparison: All Participants With Complete Usuable Data; This analysis is a comparison between the escitalopram and citalopram medication periods; Test type: Superiority or Other; p = 0.0000162, Mixed Models Analysis

3. Secondary Outcome: Number of Voxels Showing Greater Activation Following Citalopram Compared With Placebo When Affective Faces Are Presented in a Covert Stimulus Presentation and Contrasted With a Fixation Stimulus.
Description: Activation was measured using BOLD fMRI in response to affective (happy and fearful) faces presented in a covert or masked presentation and contrasted with activation in response to a neutral fixation stimulus. The response following two weeks of citalopram was compared to the response following two weeks of placebo. The cluster of differential activation was located in the right occipital fusiform gyrus.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Number; unit: voxels
Arm/Group | All Participants With Complete Usable Data
Number analyzed (Participants) | 9
voxels | 658
Statistical Analysis 1: Comparison: All Participants With Complete Usable Data; This analysis is a comparison between the citalopram and placebo medication periods; Test type: Superiority or Other; p = 0.00000936, Mixed Models Analysis

4. Secondary Outcome: Number of Voxels Showing Greater Activation Following Citalopram Compared With Placebo When Affective Faces Are Presented in a Covert Stimulus Presentation and Contrasted With a Fixation Stimulus.
Description: Activation was measured using BOLD fMRI in response to affective (happy and fearful) faces presented in a covert or masked presentation and contrasted with activation in response to a neutral fixation stimulus. The response following two weeks of citalopram was compared to the response following two weeks of placebo. The cluster of differential activation was located in the right lateral occipital cortex.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Number; unit: voxels
Arm/Group | All Participants With Complete Usable Data
Number analyzed (Participants) | 9
voxels | 253
Statistical Analysis 1: Comparison: All Participants With Complete Usable Data; This analysis is a comparison between the citalopram and placebo medication periods; Test type: Superiority or Other; p = 0.0279, Mixed Models Analysis

5. Secondary Outcome: Number of Voxels Showing Greater Activation Following Escitalopram Compared With Placebo When Affective Faces Are Presented in a Covert Stimulus Presentation and Contrasted With a Fixation Stimulus.
Description: Activation was measured using BOLD fMRI in response to affective (happy and fearful) faces presented in a covert or masked presentation and contrasted with activation in response to a neutral fixation stimulus. The response following two weeks of escitalopram was compared to the response following two weeks of placebo. The cluster of differential activation was located in the right inferior lateral occipital cortex.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Number; unit: voxels
Arm/Group | All Participants With Complete Usable Data
Number analyzed (Participants) | 9
voxels | 396
Statistical Analysis 1: Comparison: All Participants With Complete Usable Data; This analysis is a comparison between the escitalopram and placebo medication periods; Test type: Superiority or Other; p = 0.00124, Mixed Models Analysis

6. Secondary Outcome: Number of Voxels Showing Greater Activation Following Placebo Compared With Citalopram When Affective Words Are Contrasted With a Fixation Stimulus.
Description: Activation was measured using BOLD fMRI in response to affective words contrasted with activation in response to a neutral fixation stimulus. The response following two weeks of placebo was compared to the response following two weeks of citalopram. The cluster of differential activation was located in the right lingual gyrus and right superior lateral occipital cortex.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Number; unit: voxels
Arm/Group | All Participants With Complete Usable Data
Number analyzed (Participants) | 10
voxels | 619
Statistical Analysis 1: Comparison: All Participants With Complete Usable Data; This analysis is a comparison between the placebo and citalopram medication periods; Test type: Superiority or Other; p = 0.0000633, Mixed Models Analysis

7. Secondary Outcome: Number of Voxels Showing Greater Activation Following Escitalopram Compared With Citalopram When Affective Words Are Contrasted With a Fixation Stimulus.
Description: Activation was measured using BOLD fMRI in response to affective words contrasted with activation in response to a neutral fixation stimulus. The response following two weeks of escitalopram was compared to the response following two weeks of citalopram. The cluster of differential activation was located in the left primary visual cortex.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Number; unit: voxels
Arm/Group | All Participants With Complete Usable Data
Number analyzed (Participants) | 10
voxels | 289
Statistical Analysis 1: Comparison: All Participants With Complete Usable Data; This analysis is a comparison between the escitalopram and citalopram medication periods; Test type: Superiority or Other; p = 0.0241, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning with the date of the screening visit and ending with the final study visit. The average time period was approximately 4 months but varied due to differences in the length of the screening period.
Groups:
- Escitalopram: Includes all subjects who received escitalopram in one of the three medication periods
- Citalopram: Includes all subjects who received citalopram in one of the three medication periods
- Placebo: Includes all subjects who received placebo in one of the three medication periods
Arm/Group | Escitalopram | Citalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/22 | 1/21 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=22) | Citalopram (N=21) | Placebo (N=21)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
nausea (General disorders) | 1 (1) | 0 (0) | 0 (0)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Data from several subjects had to be excluded due to one or more fMRI scans with poor data quality (usually high motion) or scheduling problems that prevented a scan from occuring during the specified time window.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No